## atlas: An Interactive Text Messaging Program Combining Weather Alerts With Hyper-Localized Resources & Actionable Insights for Addressing Climate Change NCT06995755

Unique Protocol ID: R43ES035344 April 18, 2025

## Statistical Analysis Plan

This study involves a single-group, pre-post design. The primary outcome, response efficacy for taking steps to combat climate change, is assessed at individual, collective, and governmental levels from pretest (baseline) to posttest (30-day follow-up) using paired t-tests. Cohen's d will be used to report effect size as an assessment of the meaningfulness of the differences.